CLINICAL TRIAL: NCT07276529
Title: Safety and Device Functionality of the Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating Ileo-colic, Colo-colonic and Colorectal Anastomoses in Patients Undergoing Surgical Procedures
Brief Title: Initial Safety of SFM Plus OTOLoc for Creating Side-to-side or End-to-side Colorectal Anastomoses
Acronym: Colonic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-004
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Diverticular Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Diverticular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Flexagon SFM plus OTOLoc for Magnet Colon Anastomosis (Experimental): Patients will receive the Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating side-to-side Ileo-colic, Colo-colonic and side-to-side or end-to-side Colorectal Anastomoses in Patients Undergoing Surgical Procedures via endoscopic or laparoscopic delivery methods
  Interventions: Device: Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating side-to-side Colon Anatomoses

INTERVENTIONS:
Device: Flexagon Self Forming Magnet Anastomosis Plus OTOLoc for Creating side-to-side Colon Anatomoses — The SFM plus OTOLoc is used to create an immediate flow compression anastomosis for patients undergoing: Right or Left Hemicolectomy, Sigmoidectomy and Low Anterior resection

SUMMARY:
The primary objective of this trial is to investigate the safety and effectiveness of the Flexagon 25mm SFM system plus OTOLoc when used to create a side-to-side Ileo-colic, Colo-colonic and side-to-side or end-to-side colorectal anastomoses in participants undergoing colon surgery. This will be evaluated via a composite safety/effectiveness endpoint of patient success defined as successful creation of the target anastomosis without placement procedure, device or target anastomosis related reoperation through 30 days.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, early feasibility clinical study.

Patients who are scheduled for laparoscopic colon surgery requiring an anastomosis will be evaluated for participation in the study.

Study Cohorts:

* Roll-In (Training) Cohort: A roll-in phase will be included for centers that do not have previous experience with the SFM device. A maximum of 3 roll-in participants will be enrolled. Data from roll-in participants will be summarized separately from the Primary Analysis Cohort.
* Primary Analysis Cohort: A minimum of 17 participants undergoing side-to-side Ileo-colic, Colo-colonic and side-to-side or end-to-side colorectal anastomoses with the Flexagon 25mm SFM system plus OTOLoc.

Patients providing informed consent and meeting all eligibility criteria will be scheduled for surgery. All operations will be conducted by experienced general surgeons and gastroenterologists trained in the use of the Flexagon SFM System plus OTOLoc and procedures will be performed under general anesthesia.

Clinical follow-up for all participants will occur at Discharge, Day 7, 30, and 60.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22 years or older at screening
2. Candidate for surgery requiring Right of Left Hemicolectomy or Sigmoidectomy or Low Anterior resection with cardiac/medical clearance for surgery
3. Able to understand and sign informed consent document
4. American Society of Anesthesiologists (ASA) score < IV at time of procedure
5. All cancer patients must have completed chemotherapy ≥2 months prior to procedure
6. Lives, and intends to remain, within a 150-mile radius of study center for the duration of the study
7. Able to refrain from smoking during study follow-up period

Exclusion Criteria:

1. Known or suspected allergy to silicone, nickel, titanium or Nitinol
2. BMI > 55 kg/m2
3. Uncontrolled diabetes (defined as HbA1c >10%)
4. Congenital or acquired anomalies of the GI tract, including atresia or malrotation that would inhibit passing of SFM magnet
5. Participants with an acute diagnosis of obstructed or perforated colon cancer at the time of the Screening Visit
6. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous failed endoscopy that may suggest difficulty during endoscopic delivery of magnets
7. History of recurrent small bowel obstructions.
8. Coagulation deficiency not normalized by medical treatment or platelet count <50,000/µL
9. Known moderate to severe renal disease (eGFR < 44 milliliters per minute per 1.73m2) or ongoing dialysis
10. Hyperkalemia / hypercoagulability or prior Venus Thromboembolism / Pulmonary Embolism
11. Immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e., 20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents
12. Congestive heart failure with ejection fraction <35% or clinically significant arrhythmia (any rhythm disturbances except sinus tachycardia, sinus bradycardia or a sinus rhythm with premature atrial or ventricular complexes)
13. Decompensated chronic obstructive lung disease
14. Active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound.
15. Contraindication to general anesthesia
16. Breast-feeding, pregnant, or planning on becoming pregnant during the follow-up period
17. Currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent
18. Contraindication to general anesthesia
19. Participant is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Successful anastomosis created with the Flexagon SFM plus OTOLoc without reoperation. | 30 days
  The study's primary endpoint (patient success) is defined as successful anastomosis created with the Flexagon SFM plus OTOLoc without placement procedure, device or target anastomosis-related reoperation through 30 days.
Anastomosis success | 30 days
  is defined as creation of the target anastomosis without need for conversion to open procedure due to inability to create the magnet anastomosis using laparoscopic methods, intraoperative rescue procedure such as stapled or hand-sewed rescue of failed Flexagon SFM placement (i.e. - no magnet anastomosis created in patient) or intraoperative repair of adjacent organ

SECONDARY OUTCOMES:
No Bleeding at anastomosis | 30 days
  Bleeding Events through 30 days, defined as a target anastomosis related bleeding at the Flexagon SFM placement site requiring transfusion or re-operation.
No Leaks at anastomosis | 30 days
  Flexagon SFM anastomosis Leak Events through 30 days, as defined by postoperative upper GI or CT evaluation with findings consistent with anastomosis leak, or re-operative findings consistent with anastomosis leak at the Flexagon SFM placement site
No Obstructions at the anastomosis | 30 days
  Obstruction Events through 30 days as defined by the need for reintervention (e.g., endoscopic opening) or re-operation resulting from Flexagon SFM placement

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wilson, MD, Study Chair — Chief Medical Officer
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No